CLINICAL TRIAL: NCT00099151
Title: Metabolic Adaptations to Six Month Caloric Restriction
Brief Title: CALERIE (PBRC, Baton Rouge) - Comprehensive Assessment of Long-Term Effects of Reducing Intake of Energy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG0005; 5U01AG020478-02 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2004-12

CONDITIONS: Aging; Cardiovascular Disease; Diabetes Mellitus
Keywords: Longevity; Dietary restriction; Physical activity; Weight Loss; Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Motor Activity; Weight Loss | interventions — Caloric Restriction; Exercise

INTERVENTIONS:
Behavioral: Caloric Restriction (CR)
Behavioral: Exercise

SUMMARY:
This study is one of three CALERIE trials that test the hypothesis that a reduced calorie, nutritionally sound diet improves biomarkers of aging and prevents some age-related chronic diseases such as cancer, diabetes, and cardiovascular disease. The three sites that are participating in the CALERIE trial represent a diversity of subject populations and interventional strategies.

DETAILED DESCRIPTION:
This study tests whether chronic caloric restriction improves risk factors of longevity in humans as it is known to do in animals, by measuring a variety of factors dealing with metabolism and oxidative stress, through physical evaluations and laboratory tests.

Participants will receive dietary counseling and free medical evaluations. In addition, each volunteer will be asked to do one of the following:

1. Follow a reduced calorie diet
2. Follow a reduced calorie diet using a liquid diet
3. Increase physical activity while on a reduced calorie diet
4. Follow a standard diet.

Three separate five-day inpatient stays are required.

ELIGIBILITY:
Inclusion Criteria:

* Resident of greater Baton Rouge area for 1 year or longer
* Men between ages 25-50
* Women between ages 25-45
* Body Mass Index (BMI) between 25-30 (never having had BMI greater than 32)
* Healthy, non-smokers with no history of cardiovascular disease, high blood pressure, diabetes, eating disorder, or major psychiatric disorder

Exclusion Criteria:

* Pregnant or breastfeeding
* Personal history of cardiovascular disease or elevated high blood pressure (higher than 160/90 mmHg)
* Abnormal electrocardiogram (EKG)
* Personal history of diabetes
* Personal history of major psychiatric disorders
* Personal history of eating disorder
* Smoking
* Exercising regularly (more than twice a week)
* Individuals with alcoholism or other substance abuse
* Post obese (never have had a BMI greater than 32)
* Regular use of medications, except oral contraceptives
* Individuals who were ever injured by a metallic foreign body which was not removed
* Individuals who wear braces on their teeth, have non-removable false teeth, or non-removable bridgework
* Individuals in occupations requiring full alertness and motor skills (airline pilots, etc.) where even a small chance of postural dizziness would be unacceptable.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2002-03; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, Ph.D., Principal Investigator — Pennington Biomedical Research Center; Donald Williamson, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, 6400 Perkins Road, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Heilbronn LK, Ravussin E. Calorie restriction and aging: review of the literature and implications for studies in humans. Am J Clin Nutr. 2003 Sep;78(3):361-9. doi: 10.1093/ajcn/78.3.361. PMID 12936916
- [Background] Jenkins RR, Goldfarb A. Introduction: oxidant stress, aging, and exercise. Med Sci Sports Exerc. 1993 Feb;25(2):210-2. PMID 8450723
- [Background] Sohal RS, Weindruch R. Oxidative stress, caloric restriction, and aging. Science. 1996 Jul 5;273(5271):59-63. doi: 10.1126/science.273.5271.59. PMID 8658196
- [Background] Ryan AS. Insulin resistance with aging: effects of diet and exercise. Sports Med. 2000 Nov;30(5):327-46. doi: 10.2165/00007256-200030050-00002. PMID 11103847
- [Background] Masoro EJ. Food restriction in rodents: an evaluation of its role in the study of aging. J Gerontol. 1988 May;43(3):B59-64. doi: 10.1093/geronj/43.3.b59. No abstract available. PMID 3283209
- [Result] Heilbronn LK, de Jonge L, Frisard MI, DeLany JP, Larson-Meyer DE, Rood J, Nguyen T, Martin CK, Volaufova J, Most MM, Greenway FL, Smith SR, Deutsch WA, Williamson DA, Ravussin E; Pennington CALERIE Team. Effect of 6-month calorie restriction on biomarkers of longevity, metabolic adaptation, and oxidative stress in overweight individuals: a randomized controlled trial. JAMA. 2006 Apr 5;295(13):1539-48. doi: 10.1001/jama.295.13.1539. PMID 16595757
- [Derived] Allaf M, Elghazaly H, Mohamed OG, Fareen MFK, Zaman S, Salmasi AM, Tsilidis K, Dehghan A. Intermittent fasting for the prevention of cardiovascular disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013496. doi: 10.1002/14651858.CD013496.pub2. PMID 33512717
- [Derived] Thomas DM, Martin CK, Redman LM, Heymsfield SB, Lettieri S, Levine JA, Bouchard C, Schoeller DA. Effect of dietary adherence on the body weight plateau: a mathematical model incorporating intermittent compliance with energy intake prescription. Am J Clin Nutr. 2014 Sep;100(3):787-95. doi: 10.3945/ajcn.113.079822. Epub 2014 Jul 30. PMID 25080458
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151
- [Derived] Tam CS, Frost EA, Xie W, Rood J, Ravussin E, Redman LM; Pennington CALERIE Team. No effect of caloric restriction on salivary cortisol levels in overweight men and women. Metabolism. 2014 Feb;63(2):194-8. doi: 10.1016/j.metabol.2013.10.007. Epub 2013 Oct 24. PMID 24268369
- [Derived] Huffman KM, Redman LM, Landerman LR, Pieper CF, Stevens RD, Muehlbauer MJ, Wenner BR, Bain JR, Kraus VB, Newgard CB, Ravussin E, Kraus WE. Caloric restriction alters the metabolic response to a mixed-meal: results from a randomized, controlled trial. PLoS One. 2012;7(4):e28190. doi: 10.1371/journal.pone.0028190. Epub 2012 Apr 16. PMID 22523532
- [Derived] Racette SB, Das SK, Bhapkar M, Hadley EC, Roberts SB, Ravussin E, Pieper C, DeLany JP, Kraus WE, Rochon J, Redman LM; CALERIE Study Group. Approaches for quantifying energy intake and %calorie restriction during calorie restriction interventions in humans: the multicenter CALERIE study. Am J Physiol Endocrinol Metab. 2012 Feb 15;302(4):E441-8. doi: 10.1152/ajpendo.00290.2011. Epub 2011 Nov 29. PMID 22127229
- [Derived] Lecoultre V, Ravussin E, Redman LM. The fall in leptin concentration is a major determinant of the metabolic adaptation induced by caloric restriction independently of the changes in leptin circadian rhythms. J Clin Endocrinol Metab. 2011 Sep;96(9):E1512-6. doi: 10.1210/jc.2011-1286. Epub 2011 Jul 21. PMID 21778216
- [Derived] de Jonge L, Moreira EA, Martin CK, Ravussin E; Pennington CALERIE Team. Impact of 6-month caloric restriction on autonomic nervous system activity in healthy, overweight, individuals. Obesity (Silver Spring). 2010 Feb;18(2):414-6. doi: 10.1038/oby.2009.408. Epub 2009 Nov 12. PMID 19910943
- [Derived] Redman LM, Veldhuis JD, Rood J, Smith SR, Williamson D, Ravussin E; Pennington CALERIE Team. The effect of caloric restriction interventions on growth hormone secretion in nonobese men and women. Aging Cell. 2010 Feb;9(1):32-9. doi: 10.1111/j.1474-9726.2009.00530.x. Epub 2009 Oct 30. PMID 19878147
- [Derived] Anton SD, Han H, York E, Martin CK, Ravussin E, Williamson DA. Effect of calorie restriction on subjective ratings of appetite. J Hum Nutr Diet. 2009 Apr;22(2):141-7. doi: 10.1111/j.1365-277X.2008.00943.x. PMID 19302119
- [Derived] Redman LM, Heilbronn LK, Martin CK, de Jonge L, Williamson DA, Delany JP, Ravussin E; Pennington CALERIE Team. Metabolic and behavioral compensations in response to caloric restriction: implications for the maintenance of weight loss. PLoS One. 2009;4(2):e4377. doi: 10.1371/journal.pone.0004377. Epub 2009 Feb 9. PMID 19198647
- [Derived] Redman LM, Rood J, Anton SD, Champagne C, Smith SR, Ravussin E; Pennington Comprehensive Assessment of Long-Term Effects of Reducing Intake of Energy (CALERIE) Research Team. Calorie restriction and bone health in young, overweight individuals. Arch Intern Med. 2008 Sep 22;168(17):1859-66. doi: 10.1001/archinte.168.17.1859. PMID 18809812
- [Derived] Redman LM, Heilbronn LK, Martin CK, Alfonso A, Smith SR, Ravussin E; Pennington CALERIE Team. Effect of calorie restriction with or without exercise on body composition and fat distribution. J Clin Endocrinol Metab. 2007 Mar;92(3):865-72. doi: 10.1210/jc.2006-2184. Epub 2007 Jan 2. PMID 17200169
- See also: CALERIE - PBRC website — http://calerie.pbrc.edu/